CLINICAL TRIAL: NCT01403766
Title: Comparison of Estimated GFR Using Cystatin C Versus Creatinine in Pediatric Renal Transplant Patients
Brief Title: Comparison of Markers of Kidney Function
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Gentian (Unknown)
Responsible Party: Sponsor
Other Study IDs: Gentian-Cystatin-UCLA
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Chronic Kidney Disease; Renal Insufficiency
Keywords: pediatric; kidney; transplant; GFR; creatinine; cystatin C; iohexol
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric post-kidney transplant: Patients having standard of care surviellance biopsies.

SUMMARY:
Glomerular filtration rate (GFR) is the best known measurement of kidney function. Serum creatinine (blood test) is the most commonly used marker to predict GFR. It is a convenient, inexpensive test that involves a single blood draw with rapid results. However, creatinine has several limitations because its blood level is dependent on age, body mass, and sex. One of the gold standards for measuring GFR is plasma clearance of an IV injected agent, iohexol. It has been found to be safe and nontoxic in prior studies, but is not practical in the clinical setting due to the need for several timed blood draws. Recent studies have investigated the use of cystatin C as an alternative marker to predict GFR. Cystatin C also involves only a single blood draw, and has less confounding factors than creatinine since it is independent of age, body mass, and sex. Currently, it remains controversial whether cystatin C is a significantly better biomarker of estimated GFR than creatinine. To date, there has not been a large prospective cohort study to compare cystatin C and creatinine in pediatric kidney transplant patients who are on maintenance immunosuppression (anti-rejection drugs). Accurate measurement and early detection of deterioration of GFR is critical in the care of this patient population. The purpose of this study is to assess the accuracy of estimating GFR by using cystatin C versus creatinine clearance equations when compared to the surrogate gold standard of iohexol GFR in pediatric renal transplant patients.

DETAILED DESCRIPTION:
Study patients will come in for their surveillance biopsy done as standard of care post-transplant. They we be made NPO at midnight prior to the biopsy per routine. On arrival, they will have standard of care pre-biopsy bloods drawn along with baseline study labs including serum enzymatic creatinine (1mL of blood), cystatin C (1.5 mL of blood), and 1mL of blood collected pre-iohexol infusion. Two IV's will be started, one for iohexol administration and fluids, and the other for blood draws. Study patients will be started on 1x maintenance intravenous fluids. The patient will then have their standard of care protocol biopsy in the ultrasound suite. After the biopsy 5 mL Iohexol (Omnipaque 300) will be administered over 1-2 minutes, with epinephrine, solumedrol, and diphenhydramine on hand in the event of a reaction although this is very unlikely. The patient will be observed and vital signs will be taken 10 minutes post-infusion. After biopsy, maintenance fluids will be continued until completion of the study. Blood for determination of Iohexol levels (1mL) will be drawn at 10, 30, 120, and 300 minutes post iohexol infusion when patient is being observed post biopsy. At completion of the study at 300 minutes post iohexol infusion, serum creatinine (1mL of blood), cystatin C (1.5 mL of blood) will be drawn again. The total volume of blood drawn for the study will be 10mL.

Creatinine (enzymatic method) will be determined on the Olympus system, and Cystatin C (Gentian assay) will be determined on the AU400 Olympus System at the UCLA Department of Pathology and Laboratory Medicine Outreach Laboratory. Iohexol GFR will be determined at the University of Rochester Medical Center in Dr. Schwartz's laboratory. Kidney biopsies will be graded by updated Banff criteria, and reviewed by blinded pathologist.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant patient aged 1 to <19 years old
* Stable allograft function (no history of biopsy proven acute rejection or increase of creatinine of > 10% from baseline in the past 6 months)
* No changes in maintenance immunosuppression in the month before the protocol biopsy
* Subject and/or parent must be able to understand and provide informed consent

Exclusion Criteria:

* Biopsy proven acute rejection in the past 6 months
* Change in maintenance immunosuppression in the month before the protocol biopsy
* Known diabetes mellitus
* Known thyroid dysfunction
* Allergy to Iohexol or other contrast media
* Inability or unwillingness of a participant or their legal guardian to give written informed consent or comply with the study protocol

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will be recruited from UCLA pediatric kidney transplant patients with stable allograft function that come in for routine surveillance biopsy. Patients will be induced with either daclizumab, basiliximab, or thymoglobulin and maintained on tacrolimus, mycophenolate mofetil, and steroid-free or steroid-based immunosuppression.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is a comparison of determination of GFR through three methods: cystatin C (Gentian assay), creatinine (Schwartz and update Schwartz) and iohexol disappearance | Participants will be followed for the duration of the Iohexol GFR measurement (approximately 8 hours) that will take place at the time of surveillance biopsy at either 6 months, 1 or 2 years post-transplant..

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States